CLINICAL TRIAL: NCT02931877
Title: Comparison of Postoperative Outcome and Cognitive Function After Sevoflurane and Propofol Anaesthesia for Cardiac Valvular Surgery With Cardiopulmonary Bypass
Brief Title: Comparison of Postoperative Outcome After Sevoflurane and Propofol Anaesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Hong Li, Director, Department of Anesthesiology, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Li Hong-Group
Record Dates: First submitted 2016-10-10; First posted 2016-10-13 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Sevoflurane; Propofol; Cardiac valvular surgery; Cardiopulmonary bypass; Postoperative cognitive dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sevoflurane (Experimental): Maintenance of anesthesia with sevoflurane during the cardiac valvular surgery.
  Interventions: Drug: sevoflurane
- Propofol (Active Comparator): Maintenance of anesthesia propofol during the cardiac valvular surgery.
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: sevoflurane
  Arms: Sevoflurane
Drug: propofol
  Arms: Propofol

SUMMARY:
As the investigators know, postoperative cognitive dysfunction (POCD) is a fairly well-documented clinical phenomenon, which affect patients' short-term and long-term outcome. Most patients will receive general anesthesia and cardiopulmonary bypass (CPB) during cardiac valvular surgery. Inhalation sevoflurane based and propofol based anesthesia are most commonly used strategy for general anesthesia. At present, it was unknown that which one is better in providing cerebral protection effect for patients undergoing cardiac valvular surgery with CPB. The current study aimed to explore the possible difference.

DETAILED DESCRIPTION:
The investigators hypothesize that the incidence of postoperative cognitive dysfunction (POCD) is not different in patients received intravenous anesthetics propofol or sevoflurane for their cardiac valvular surgery. Two groups of general anesthetics (propofol or sevoflurane) are used to explore the possible difference of the postoperative outcome and the incidence of POCD. After cardiac valvular surgery with CPB, patients' POCD tests at 7 days after the surgery, and postoperative delirium, etc., are evaluated by different questionnaires. Also the blood sample of these patients are collected for detection of some stress hormones.

ELIGIBILITY:
Inclusion Criteria:

* patients who receive cardiac valvular surgery
* 18 to 65 years
* American society of anesthesiologists classification Ⅱto Ⅲ
* education level higher than elementary school

Exclusion Criteria:

* Patients are not expected to be alive for longer than 3 months.
* Mini-mental State Examination (MMSE) score ≤ 23.
* current use of sedatives or antidepressant
* history of dementia, psychiatric illness or any diseases of central nervous system.
* accompanying liver or kidney function deficiency
* history of some endocrine disease
* alcoholism and drug dependence
* patients previously included in this study or currently included in the other clinical study
* patients who have second surgery during the study period
* difficult to follow up or patients with poor compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with postoperative cognitive dysfunction (POCD) | From 7 days after the surgery to the day of discharge from hospital
  POCD is a composite outcome measure

SECONDARY OUTCOMES:
Postoperative delirium (POD) | Up to 7 days after the surgery
  POD is evaluated by a commonly used questionnaire

OTHER OUTCOMES:
Degree of increase of stress hormones | Up to 24 hours after the surgery
  Stress hormones include S-100β, Il-6, etc.
Length of ICU stay | Up to 7 days after the surgery
  The time for patient stay in ICU
Length of hospital stay | Up to 3 months after the surgery
  The time for patient stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Hong Li, M.D., Principal Investigator — Department of Anesthesiology, Xinqiao Hospital, Third Military Medical University
Locations (3):
- China (3):
  - Xinan Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Xinqiao Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality

IPD SHARING:
Plan to Share IPD: Undecided